CLINICAL TRIAL: NCT06751381
Title: A Prospective Study on Monitoring Salivary Gland Injury in Nasopharyngeal Carcinoma Patients After Radiotherapy Using Multi-Modal Radiomics
Brief Title: Monitoring Salivary Gland Injury in Nasopharyngeal Carcinoma Patients After Radiotherapy Using Multi-Modal Radiomics
Status: Not yet recruiting | Type: Observational
Sponsor: Hainan Medical College (Other)
Responsible Party: Principal Investigator, Shui Bin Juan, Principal Investigator (Graduate Research), Hainan People's Hospital
Other Study IDs: ShuiBinJuan-2024-NPC001
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Nasopharyngeal Carcinoma ,Xerostomia,Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Nasopharyngeal Carcinoma Patients
  Interventions: Device: IVIM Imaging MRF Imaging

INTERVENTIONS:
Device: IVIM Imaging MRF Imaging — IVIM imaging will be performed to evaluate microstructural and perfusion changes in the salivary glands of nasopharyngeal carcinoma patients undergoing radiotherapy. This technique quantifies diffusion and perfusion parameters, providing insights into early tissue damage.
  MRF imaging will be used to quantify salivary gland tissue characteristics, including relaxation parameters (T1 and T2 mapping), to monitor radiotherapy-induced damage. The technique enables precise tissue characterization through multi-parametric MRI.

SUMMARY:
This prospective observational study aims to evaluate the role of intravoxel incoherent motion (IVIM) imaging and magnetic resonance fingerprinting (MRF) techniques in monitoring salivary gland injury in nasopharyngeal carcinoma (NPC) patients undergoing radiotherapy. The study will recruit patients diagnosed with NPC who are receiving standard radiotherapy, and quantitative imaging data will be collected using IVIM and MRF techniques at multiple time points, including pre-treatment, during radiotherapy, and post-treatment. The primary objective is to analyze changes in salivary gland structure and function and to identify early imaging biomarkers indicative of radiation-induced injury. The findings are expected to provide new insights into the dynamic progression of salivary gland damage, establish predictive models for the risk of xerostomia, and guide the development of personalized therapeutic strategies to mitigate long-term complications.

DETAILED DESCRIPTION:
This is a prospective study designed to investigate the application of intravoxel incoherent motion (IVIM) and magnetic resonance fingerprinting (MRF) imaging techniques in monitoring salivary gland injury in nasopharyngeal carcinoma (NPC) patients after radiotherapy. The study aims to quantify and assess salivary gland function changes during and after radiotherapy using advanced imaging technologies, with the goal of identifying early imaging biomarkers associated with radiation-induced damage.

Patients diagnosed with NPC and receiving standard radiotherapy will be recruited. Imaging data will be acquired at three time points: prior to radiotherapy (baseline), during radiotherapy (mid-course), and after radiotherapy (post-treatment). IVIM and MRF sequences will be performed to collect data on salivary gland microstructure, perfusion, and relaxation properties. These parameters will be analyzed to detect early changes in salivary gland function and correlate them with the development of xerostomia.

This study is expected to provide valuable insights into the utility of IVIM and MRF imaging in predicting and monitoring radiation-induced salivary gland damage. The findings may facilitate early intervention strategies and contribute to personalized radiotherapy planning aimed at minimizing xerostomia risk in NPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of nasopharyngeal carcinoma.
2. Scheduled to undergo radiotherapy as part of standard treatment.
3. Aged 18 years or older.
4. No contraindications to MRI scans (e.g., no implanted metallic devices).
5. Written informed consent has been provided.

Exclusion Criteria:

1. Contraindications to MRI, such as metallic implants or claustrophobia.
2. Severe comorbid conditions, including significant renal or hepatic dysfunction.
3. Concurrent participation in another interventional clinical trial.
4. Pregnant or breastfeeding.
5. Any condition that may impair compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18 years or older) with a confirmed diagnosis of nasopharyngeal carcinoma who are scheduled to undergo radiotherapy as part of standard treatment. Recruitment will occur at the Department of Radiotherapy, Hainan Provincial People's Hospital. Eligibility requires the ability to undergo MRI scans and the provision of informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure • Title: Quantitative assessment of salivary gland changes using IVIM and MRF imaging • Time Frame: From baseline to 6 months post-radiotherapy • Description: Quantification of salivary gland microstructural, perfusion, and re | From baseline to 6 months post-radiotherapy
  IVIM Imaging: Quantification of salivary gland microstructural and perfusion changes using IVIM-derived parameters (D, D*, f values) to evaluate radiotherapy-induced changes.
  MRF Imaging: Quantification of salivary gland relaxation properties using MRF-derived relaxation times (T1 and T2 mapping) to evaluate radiotherapy-induced changes.
  Unit of Measure:
  IVIM: D, D*, f values MRF: T1 and T2 relaxation times Analysis: Changes in salivary gland microstructure and perfusion (IVIM parameters) as well as relaxation properties (MRF parameters) will be assessed separately from baseline to 6 months post-radiotherapy.

IPD SHARING:
Plan to Share IPD: No